CLINICAL TRIAL: NCT00174031
Title: Prevalence and Profiles of Sports Injury in Taiwanese Adolescent Baseball Players
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701434
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 1993-09

CONDITIONS: Sports Injury
Keywords: baseball; injury
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To investigate prevalence and profile of sports injury in Taiwanese adolescent baseball players in a longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese adolescent baseball players

Exclusion Criteria:

* Who are not willing to join this study

Ages: 10 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800
Dates: Start 1993-12

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Director — School and Graduate institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, NTU, Taiwan, Taipei, Taiwan